CLINICAL TRIAL: NCT01524432
Title: Phase III Study in Hygienic Socks With Antifungal Agent-loaded Microcapsules for Patients With Tinea Pedis
Brief Title: Hygienic Socks With Antifungal Agent-loaded Microcapsules for Patients With Tinea Pedis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prof. Yuen Chun-Wah (Other)
Collaborators: Dr. Cheung Hing Cheong Private Dermatology Clinic (Unknown)
Responsible Party: Sponsor-Investigator, Prof. Yuen Chun-Wah, Professor, The Hong Kong Polytechnic University
Organization: The Hong Kong Polytechnic University (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Mic_Clo_Terb
Record Dates: First submitted 2012-01-18; First posted 2012-02-02 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2013-03

CONDITIONS: Tinea Pedis
Keywords: Clotrimazole; Microcapsules
MeSH Terms: conditions — Tinea Pedis | interventions — Clotrimazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug loaded microcapsules socks (Experimental): Study medication
  Interventions: Drug: Anti-fungal agent (Clotrimazole) loaded microcapsules
- No drug loaded microcapsules socks (Placebo Comparator): Placebo medication
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anti-fungal agent (Clotrimazole) loaded microcapsules — Clotrimazole loaded microcapsules padded on socks and the patient should wear the socks every day for 2 weeks
  Other Names: Anti-fungal agent loaded microcapsules
  Arms: Drug loaded microcapsules socks
Drug: Placebo — No drug loaded microcapsules socks
  Arms: No drug loaded microcapsules socks

SUMMARY:
This is a study of hygienic socks with antifungal agent-loaded microcapsules for subjects with interdigital type tinea pedis (athlete's foot between the toes). This is a 6 week study which has a 2 week treatment period and a 4 week follow-up evaluation.

DETAILED DESCRIPTION:
Tinea pedis (Athlete's Foot) is a common skin disease which affects a large number of the population. The development of hygienic socks through the microencapsulation technology have great potential to provide the convenient pharmacological treatment on one hand, and good moisture management which can reduce the microbial overgrowth on the other hand for patients with tinea pedis. The socks, therefore, reduce the effects of the skin disease on the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age and of either sex.
* Subjects must have clinical evidence of interdigital tinea pedis of one or both feet characterized by: (i) moderate erythema, (ii) scaling and (iii) mild pruritis.
* Have microscopic evidence (positive KOH) of the presence of fungi. Evaluable subjects must have a positive KOH and a fungal culture positive for a dermatophyte in the skin scrapings taken at the Baseline Visit. Subjects with a positive KOH may be entered into the study pending the results of the fungal culture
* Be willing and able to give informed consent/assent or have their parent/guardian do so, if applicable.
* Be willing and able to use the assigned study medication as directed and to commit to all follow-up visits for the duration of the study.
* Be in good health and free of any disease or physical condition which might, in the Investigator's opinion, expose the subject to an unacceptable risk by study participation.
* Females must be non-pregnant, non-lactating and not intending to become pregnant during the course of the study.

Exclusion Criteria:

* Is pregnant, nursing or planning a pregnancy during the study.
* Has used topical antifungals or topical corticosteroids on the feet within 4 weeks prior to the start of the study.
* Has received systemic antifungal therapy within 4 weeks prior to the start of the study medication.
* Has used systemic antibacterials or systemic corticosteroids within 4 weeks prior to the start of the study. Systemic corticosteroids do not include intranasal, inhaled, and ophthalmic corticosteroids used for the management of allergies, pulmonary disorders or other conditions.
* Has a history of uncontrolled diabetes mellitus or is immunocompromised (due to disease, e.g., HIV, or medications).
* Has concurrent tinea infection e.g. Tinea Versicolor, Tinea Cruris, Moccasin-type Tinea Pedis, etc. (in the opinion of the Investigator).
* Onychomycosis, involving ≥ 20% of the area of either great toenail or involvement of more than five toenails in total.
* Has any other skin disease which might interfere with the evaluation of tinea pedis.
* Is currently enrolled in an investigational drug or device study.
* Has received an investigational drug or treatment with an investigational device within 30 days prior to entering this study.
* Is unreliable, including subjects with a history of drug or alcohol abuse.
* Has known hypersensitivity to any of the components of the study medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
• Complete Cure | Day 44
  Complete Cure is defined as a negative KOH and negative fungal culture and no evidence of clinical disease for each sign and symptom at Day 44.

SECONDARY OUTCOMES:
Effective Treatment | Day 44
  Effective Treatment defined as negative KOH, negative fungal culture, no or mild erythema and/or scaling with all other signs or symptoms being absent at Day 44.

CONTACTS AND LOCATIONS:
Overall Officials: Chun Wah M. Yuen, Principal Investigator — Hong Kong PU
Locations (1):
- Institute of Textiles and Clothing, The Hong Kong Polytechnic University, Kowloon, Hong Kong